CLINICAL TRIAL: NCT02638974
Title: Feasibility and Acceptability of Medical Skin Camouflage for Recovery of Women With Self-Harm Scarring in Prison
Brief Title: Skin Camouflage for Women Prisoners With Self-Harm Scarring
Acronym: COVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government)
Responsible Party: Principal Investigator, Kerry Gutridge, Project Manager, University of Manchester
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15438
Record Dates: First submitted 2015-11-18; First posted 2015-12-23 (Estimated); Results first posted 2019-10-18 (Actual); Last update posted 2019-10-18 (Actual); Status verified 2019-09

CONDITIONS: Self Injurious Behaviour
MeSH Terms: conditions — Self-Injurious Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical Skin Camouflage (Experimental): This arm will use medical skin camouflage for 6 weeks
  Interventions: Other: Medical Skin Camouflage
- Wait List Control (No Intervention): This arm will receive medical skin camouflage at the end of the study

INTERVENTIONS:
Other: Medical Skin Camouflage — Medical skin camouflage is a prescription preparation designed to cover scars and other skin conditions
  Arms: Medical Skin Camouflage

SUMMARY:
Women prisoners are more likely to commit suicide or self-harm than women in the community or male prisoners.

Healthcare services have improved how they manage self-harm in the community and prisons. However, there has been little focus on the recovery of people with self-harm scars. Medical skin camouflage (MSC) is a British National Formulary-listed topical cream designed to cover skin conditions. Research on MSC has focused on its use with non-self-harm marks e.g. burns. The evidence from this research suggests that the cream helps women feel better and do more activities. There is little/no evidence about the effects of the preparation for women who self-harm and for prisoners.

This research was funded by the National Institute for Health Research Research for Patient Benefit Programme. In the research the investigators will examine whether it is possible and practical to use MSC in prison. The investigators will ask women prisoners and staff what they think about the cream. The research has four parts. In the first part the investigators will run focus groups with women prisoners and prison staff to find out the best way to deliver the MSC intervention and how to measure its effects. In the second part the investigators will design a programme for delivering the MSC. The investigators will then train 6-10 long-term prisoners to become skin camouflage practitioners. The final part will involve a small randomised controlled trial with 40 women prisoners; 20 will be allocated to the intervention group and will use the MSC for 6 weeks. The investigators will measure their mood, thoughts of self-harm and wellbeing before and after they use MSC. The investigators will compare these results with 20 women who have not used MSC (waitlist control group). All women taking part will be placed at random into the control or the treatment group. The control group will receive the MSC after the research has ended.

Potential benefits of this study may be an increase in self-esteem and quality of life for the women prisoners. As women recover they may be less likely to self-harm.

DETAILED DESCRIPTION:
The study aims to establish the feasibility and acceptability of the use of medical skin camouflage for self-harm scarring in a women's prison. The investigators are interested in the use of medical skin camouflage by women who are recovering from self-harm. The research location is a Closed Category prison for female adults and young offenders in England. The study will involve adult women prisoners (over 18) and staff at the prison.

Medical Skin Camouflage uses specialised creams/powders to disguise skin conditions or scarring with the intention of normalising the appearance of the skin. Studies which have examined the use of medical skin camouflage for dermatological diseases or burns have reported significant psychological benefits and social benefits. Preliminary findings from co-applicant Dr Sandeep Ranote's work, with young people who self-harm in the community, indicate that the use of medical skin camouflage can lead to increased well-being, confidence and ability to partake in social activities. Currently there is no evidence on the use of MSC for self-harm scarring in prisons.

The research design is intended to provide information necessary to decide whether it is feasible and acceptable to conduct a full scale randomised controlled trial of MSC in a women's prison. The four phases of the research are as follows:

Phase 1: Focus groups in prison. Interested prisoners and staff will be provided with an information sheet about phase 1 of the project and will have up to 48 hours to decide whether they want to take part in this phase of the research. After consent the investigators will conduct 2 focus groups with women prisoners (including current self-harmers) and prison staff (6-10 in each group; 12-20 in total). The focus groups are designed to achieve two aims: to ensure that appropriate outcome measures are used in the phase four pilot trial; and to explore any barriers to the delivery of medical skin camouflage in a prison environment. The focus groups will last 60-90 minutes.

In the groups the investigators shall explore the following:

1. Any potential problems with the introduction of MSC.
2. How training long-term prisoners as camouflage practitioners will be undertaken (see phase 3).
3. With women prisoners: the investigators will discuss how scarring affects mood, self-esteem, self-confidence, resilience, and how others perceive them. These questions will be designed to assess how best to collate information about how scarring affects prisoner's lives and their mental health informing which outcomes should be measured in phase 4. Part of this consultation will involve asking them to help us adapt standard measures of wellbeing (such as WEMWES) so they are appropriate for a prison environment.
4. The investigators will also discuss the use of Assessment, Care in Custody and Teamwork data (ACCT) and Inpatient Mental Health Records during the pilot trial. Prisoners who are at risk of self-harm are assessed by the prison Safer Custody team who follow the ACCT procedures which include recording incidents of self-harm.

The focus groups will be recorded, transcribed and checked for accuracy. The data will be analysed by members of the research team. To mitigate against possible researcher bias, an independent experienced researcher will review the findings.

During phase 1 members of the research team will also be trained to become medical skin camouflage practitioners. This training will be delivered by Changing Faces, a third-sector organisation. Training is accredited by the Royal College of Nursing (2012). This training will be done in preparation for phase 3.

Phase 2: Guidance protocol

Using the findings from phase 1, the investigators will refine the study processes and procedures ready for the next two phases. This will involve:

1. The production of a guidance protocol for the use of medical skin camouflage in prisons. The protocol will focus on practical aspects of where, when and how treatment is delivered, who applies it; how it is applied; how it is prescribed, and storage of prescribed products.
2. Finalising how the training of lifers will be delivered and supported (in preparation for phase 3). This includes adapting the Changing Faces training manual so it is suitable for use with women prisoners.
3. Finalising the eligibility criteria for phase 4, e.g. how assessment will be made of self-harm scar wounds and how women will be referred to the trial.
4. Finalising the outcome measures to be used in phase 4.
5. If necessary, refining our standard operating procedures for monitoring and managing any incidents of self-harm during the intervention.

Phase 3: Training lifers This phase of the research involves the training of long-term prisons (lifers) to deliver the medical skin camouflage intervention to the women prisoners in phase 4. By training lifers to deliver the intervention the investigators will ensure that women prisoners are integral to the delivery of camouflage to other women offenders. Not only does this genuinely include stakeholders in research, but it also builds sustainable capacity within the prison and is likely to increase self-efficacy/self-worth of those women.

In phase 3 the MSC trained research team members will implement a rolling programme of training and support for 6 or more long-term women prisoners so they are able to deliver the MSC intervention. During this phase and in phase 4, the research team will provide regular mentoring and advice on practical aspects of the product use. The women lifers will receive ongoing supportive liaison throughout the project from members of the research team.. The project manager will liaise with the prison lifers to ensure fidelity to the guidance protocol.

Phase 4 Phase 4 is a small scale randomised wait list control pilot. A sample of 40 women prisoners with self-harm scarring at the prison will be recruited; 20 participants will be randomised to receive the 6 week camouflage intervention; 20 participants will become wait-list controls and receive the intervention after completion of the 6-week trial. The trial participants will be remand and sentenced women prisoners screened for date of release, with at least 6 weeks left on their sentence and self-harm scarring, with closed wounds (to allow the MSC to be applied).

Eligible female prisoners will be identified by the prison, for example using information known by the Safer Custody team. Once identified the research team will provide the potential participants with an information sheet. Following earlier research in prisons, the investigators envisage that potential participants will be allocated a research number assuring anonymity from the research team. This process will allow the researchers to send out participant information sheets to relevant potential participants and allow participants to make an informed decision about participation prior to identifying themselves to researchers. Potential participants will be given 24-48 hours to decide whether they want to consent to involvement. The Clinical Research Network will assist the research assistant with the recruitment to the pilot trial.

A member of the research team will interview all the women at the start of the trial collecting information on the following:

1. Basic demographics (Bespoke Personal History Questionnaire)
2. History of self-harm (Deliberate Self-harm Inventory)
3. Mood (Beck Depression Inventory II, Beck Scale for Suicidal Ideation, Beck Hopelessness Scale)
4. Psychosocial well-being (Warwick Edinburgh Mental Wellbeing Scale) and self-esteem (Rosenberg Self-esteem Scale)
5. Health-related quality of life (SF-12 and EQ5D) and quality of life related to scarring (Prison-adapted Dermatology Quality of Life Index)
6. Zanarini Rating Scale for Borderline Personality Disorder With women's permission the research team will record key clinical characteristics from CNomis, SystemOne (the prison electronic medical records) and from ACCT documentation.

The MSC treatment will be provided for 6 weeks. The trained long-term prisoners will run regular 1 hour appointments for women in the intervention group. During this appointment, the participant will receive information about the specially formulated MSC creams. The lifers will take them through the skin tone colour-matching process and will try small amounts of cream until they find a match. After this, they will apply the cream to a larger area and use special powders to set the cream and make sure it is waterproof. Throughout the appointment, an explanation of what they are doing will be given to participants and the participant will then be able to try applying the camouflage creams themselves. When they are happy with how it looks, the practitioner will complete a prescription form that will be processed by a nurse prescriber. The prescription will provide them with one cream and one powder which we anticipate will last for 3-6 months. During the intervention the research team will record data on new self-harm incidents and related life-events (using ACCT data and Inpatient mental health records). All participants will also be asked to complete a weekly diary to record their self-harm experiences (thoughts and acts) during the trial.

At the end of the 6 weeks the research team will meet with participants to collect post intervention data. Initial post-intervention testing is at 6 weeks as the average sentence length for women in the prison. Six weeks post-intervention the investigators will repeat baseline measures apart from the demographic questionnaire. A final follow-up will be piloted at 3-months post-baseline. Recruitment, participation, retention and causes of drop-out will also be collected.

Post-intervention the investigators will conduct qualitative interviews with the following groups:

1. All women who received the intervention will be invited to participate in an interview to explore their experience of the intervention and its acceptability. The investigators will explore the participants views on treatment accessibility and potential impact on how women feel about their scarring, mood, self-esteem and self-confidence.
2. All women in the waitlist control group will be invited to participate in an interview to explore their experiences of being randomised to the control group and participating in the research.
3. 6-10 prison health and other staff who have direct contact with the participants will take part in a focus group. This will explore their views in relation to the treatments' acceptability and perceived effects on participants' well-being, quality of life and everyday functioning.
4. Interviews will be conducted with the lifers who delivered the intervention exploring how acceptable the training was, how MSC was used with the participants, feedback on the mentoring and support and any benefits or difficulties working with participants.

During the course of the research the investigators will also be exploring the best way to calculate the resource use associated with providing MSC in prisons. The investigators shall develop a bespoke resource use questionnaire to pilot the collection of resource use data concerning the delivery of the intervention, including time spent by Changing Faces training the research team, time spent by trained prisoners delivering the intervention, and quantities of MSC products used and prescribed. Descriptive analysis of this data will inform future trial design.

The Secure Facilities Service Use Schedule (SF-SUS) will be used to collect other relevant resource-use at 3month follow-up: contact with personal, Safer custody and general prison officers, and staff from mental health team; time on one-to-one observation, specialist mental health units; recording observations and care plans. SF-SUS records individual-level data on service use within secure facilities and external services for economic evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Remand and sentenced women prisoners screened for date of release with at least 6 weeks left on their sentence
* Self-harm scarring, with closed wounds (to allow the MSC to be applied).
* Able to give written, informed consent.

Exclusion Criteria:

* Women prisoners with open wounds
* Less than 6 weeks on anticipated release date
* Women with skin conditions and allergies
* Women prisoners who lack the capacity to consent to the research.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Abel, PhD, Principal Investigator — University of Manchester
Locations (1):
- Styal Prison, Wilmslow, Cheshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mitchell H, Abel KM, Dunlop BJ, Walker T, Ranote S, Robinson L, Edgar F, Millington T, Meacock R, Shaw J, Gutridge K. Acceptability and feasibility pilot randomised controlled trial of medical skin camouflage for recovery of women prisoners with self-harm scarring (COVER): the study protocol. BMJ Open. 2019 Jan 17;9(1):e021891. doi: 10.1136/bmjopen-2018-021891. PMID 30782675

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Medical Skin Camouflage | Wait List Control
Started | 26 | 25
Completed | 23 | 22
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Medical Skin Camouflage | Wait List Control | Total
Number analyzed (Participants) | 26 | 25 | 51
Age, Continuous [Mean (Full Range); unit: years] — Population: Participants withdrew from the research
  years
    number analyzed (Participants) | 23 | 23 | 46
    (all) | 31 [21 to 47] | 29 [19 to 51] | 30 [19 to 51]
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Participants withdrew from the research
  Participants
    number analyzed (Participants) | 23 | 23 | 46
    Female | 23 | 23 | 46
    Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Participants withdrew from the research
  Participants
    Ethnicity: number analyzed (Participants) | 23 | 23 | 46
    Ethnicity: White | 22 | 22 | 44
    Ethnicity: Non-white | 1 | 1 | 2
Adapted-Dermatology Quality of Life Index [Mean (Standard Deviation); unit: score on a scale] — Adapted DQLI Minimum 0, Maxium 24. The higher the score ont he DQLI, the more impaired the quality of life. Population: Participants withdrew from the study so their data was not analysed
  score on a scale
    number analyzed (Participants) | 23 | 23 | 46
    (all) | 12.6957 (3.95928) | 12.2609 (6.51723) | 12.4783 (5.33641)
Beck's Depression Inventory [Mean (Standard Deviation); unit: score on a scale] — BDI-II Minimum 0 Maximum 63. 0-13 indicates minimal depression, 14-19 mild depression, 20-28 moderate depression, 29-63 severe depression Population: Participants withdrew from the research
  score on a scale
    number analyzed (Participants) | 23 | 23 | 46
    (all) | 33.6957 (11.39950) | 38.9565 (6.99011) | 36.3261 (9.72066)
Beck's Hopelessness Scale [Mean (Standard Deviation); unit: score on a scale] — BHS Minimum 0 Maximum 20. 0-3 indicates no or minimal hopelessness, 4-8 is mild, 9-14 is moderate and 15+ is severe Population: Participants withdrew from the research.
  score on a scale
    number analyzed (Participants) | 23 | 23 | 46
    (all) | 10.0000 (5.86980) | 14.6957 (4.43575) | 12.3478 (5.66556)
Beck's Scale for Suicide Ideation [Mean (Standard Deviation); unit: score on a scale] — BSS Minimum 0 Maximum 28. The higher the score the greater the suicidal ideation. Population: Participants withdrew from the research or decline to answer this scale
  score on a scale
    number analyzed (Participants) | 22 | 22 | 44
    (all) | 6.2273 (7.75783) | 8.8636 (8.66463) | 7.5455 (8.23621)
Warwick-Edinburgh Mental Wellbeing Scale [Mean (Standard Deviation); unit: score on a scale] — WEMWBS Minimum 14 Maximum 70. Higher scores represent higher wellbeing Population: Participants withdrew from the research.
  score on a scale
    number analyzed (Participants) | 23 | 23 | 46
    (all) | 36.0435 (11.17008) | 30.2609 (9.12647) | 33.1522 (10.50072)
Rosenberg Self Esteem Scale [Mean (Standard Deviation); unit: score on a scale] — RSE Minimum 0 Maximum 30. Higher scores represent higher self esteem. Population: Participants withdrew from the research
  score on a scale
    number analyzed (Participants) | 23 | 23 | 46
    (all) | 11.6522 (4.68662) | 9.6087 (3.38095) | 10.6304 (4.17058)

OUTCOME MEASURES:

1. Primary Outcome: Warwick-Edinburgh Mental Well-being Scale
Description: WEMWBS, Minimum: 14 Maximum: 70. Higher scores represent higher mental wellbeing
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Skin Camouflage | Wait List Control
Number analyzed (Participants) | 23 | 22
score on a scale | 40.1739 (8.97295) | 30.8182 (8.46076)

2. Secondary Outcome: Becks Scale for Suicidal Ideation
Description: BSS MInimum: 0 Maximum: 28. The higher the score the greater the suicidal ideation.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Skin Camouflage | Wait List Control
Number analyzed (Participants) | 23 | 22
score on a scale | 5.0435 (10.20463) | 4.9412 (6.76822)

3. Secondary Outcome: Becks Depression Inventory
Description: BDI-II Minimum: 0 Maximum: 63. 0-13 indicates minimal depression; 14-19 mild depression; 20-28 moderate depression and 29-63 severe depression
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Skin Camouflage | Wait List Control
Number analyzed (Participants) | 23 | 22
score on a scale | 25.6957 (16.93687) | 35.1364 (8.45884)

4. Secondary Outcome: Becks Hopelessness Scale
Description: BHS, Minimum: 0 Maximum: 20. 0-3 indicates No or minimal hopelessness; 4-8 is mild; 9-14 is moderate and 15+ is severe
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Skin Camouflage | Wait List Control
Number analyzed (Participants) | 23 | 22
score on a scale | 7.3636 (5.57670) | 12.0000 (6.11010)

5. Secondary Outcome: Rosenberg Self-Esteem Scale
Description: RSE Minimum: 0 Maximum: 30 Higher scores represent higher self-esteem
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Skin Camouflage | Wait List Control
Number analyzed (Participants) | 23 | 22
score on a scale | 14.8696 (4.21366) | 12.1818 (4.39303)

6. Secondary Outcome: Adapted-DQLI
Description: Adapted-DQLI Minimum: 0 Maximum: 24 The higher the score on the Dermatology Quality of Life Index the more impaired the quality of life
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Medical Skin Camouflage | Wait List Control
Number analyzed (Participants) | 23 | 22
score on a scale | 6.7391 (5.42902) | 11.9091 (6.11718)

ADVERSE EVENTS:
Time Frame: 9 weeks
Arm/Group | Medical Skin Camouflage | Wait List Control
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 0/26 | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-01-08): https://cdn.clinicaltrials.gov/large-docs/74/NCT02638974/Prot_SAP_000.pdf